CLINICAL TRIAL: NCT00432926
Title: Behavior Change and Maintenance Intervention for HIV+ MSM Methamphetamine Users
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of California, San Diego (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Principal Investigator, Thomas L. Patterson, Principal Investigator, University of California, San Diego
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: R01DA021115 (NIH); R01DA021115 (NIH)
Record Dates: First submitted 2007-02-06; First posted 2007-02-08 (Estimated); Last update posted 2012-09-28 (Estimated); Status verified 2012-09

CONDITIONS: HIV Infections; Substance Abuse; Sexually Transmitted Diseases
Keywords: HIV; STDs; Methamphetamine abuse; MSM; HIV Seronegativity
MeSH Terms: conditions — HIV Infections; Substance-Related Disorders; Sexually Transmitted Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- 1 (Experimental): Five-session behavior change intervention that combines client-centered motivational interviewing and structured behavioral counseling (to address context of unsafe sex/drug use; condom use, safer sex negotiation; disclosure; and enhancement of social supports).
  Interventions: Behavioral: EDGE counseling, no maintenance
- 2 (Experimental): Five-session behavior change intervention (identical to Arm 1) that combines client-centered motivational interviewing and structured behavioral counseling (to address context of unsafe sex/drug use; condom use, safer sex negotiation; disclosure; and enhancement of social supports) PLUS eight group-format safer sex maintenance counseling sessions, which utilize clinical strategies from relapse prevention to identify high risk situations and develop effective coping strategies.
  Interventions: Behavioral: EDGE counseling, plus maintenance
- 3 (Active Comparator): An attention-control condition that is time-equivalent to Arm 2, and addresses diet, exercise, and HIV.
  Interventions: Behavioral: Attention control

INTERVENTIONS:
Behavioral: EDGE counseling, no maintenance — Five-session behavior change intervention that combines client-centered motivational interviewing and structured behavioral counseling (to address context of unsafe sex/drug use; condom use, safer sex negotiation; disclosure; and enhancement of social supports).
  Arms: 1
Behavioral: EDGE counseling, plus maintenance — Five-session behavior change intervention (identical to Arm 1) that combines client-centered motivational interviewing and structured behavioral counseling (to address context of unsafe sex/drug use; condom use, safer sex negotiation; disclosure; and enhancement of social supports) PLUS eight group-format safer sex maintenance counseling sessions, which utilize clinical strategies from relapse prevention to identify high risk situations and develop effective coping strategies.
  Arms: 2
Behavioral: Attention control — An attention-control condition that is time-equivalent to Arm 2, and addresses diet, exercise, and HIV.
  Arms: 3

SUMMARY:
This study tests the effectiveness of a behavioral intervention to reduce sexual risk behavior in HIV-positive, methamphetamine-using men who have sex with men (MSM). It builds on the findings of a previous study (R01 DA012116, "Promoting safer sex in HIV+ homosexual and bisexual men who use methamphetamine"). That study achieved significant short-term results that eroded over time. Accordingly, this study hypothesizes that the addition of a maintenance component to the already proven counseling and educational components of the treatment model will result in longer-lasting positive effects.

DETAILED DESCRIPTION:
Methamphetamine use by MSM has been consistently associated with increased HIV transmission. In the previous funding period we demonstrated reductions in transmission risk behavior associated with participation in our behavioral intervention; however, these improvements eroded over time, underscoring the need to develop and test interventions designed to enhance longer-term behavior change. The objective of this study is to evaluate the efficacy of an intervention designed to maintain reductions in high-risk sexual practices achieved by methamphetamine-using HIV+ MSM. Three major questions addressed are: 1) Can methamphetamine-using HIV+ MSM modify their high-risk sexual practices over an extended (16-month) period? 2) Do "group maintenance sessions" result in less erosion of behavioral improvements? 3) Are the underlying mechanisms the same for acquisition and maintenance of behavior change? We will assign 450 sexually active HIV+ MSM who regularly use methamphetamine and who have had unprotected sex with an HIV-negative or unknown-status partner to one of three conditions: 1) an eight-session intervention, combining client-centered motivational interviewing and structured behavioral counseling to address five intervention domains (context of unsafe sex/drug use; condom use; safer sex negotiation; disclosure; and enhancement of social supports); 2) the same eight counseling sessions (i.e., identical to condition 1 above), plus eight group-format safer sex maintenance sessions, which utilize clinical strategies from relapse prevention to identify high-risk situations and develop effective coping strategies; or 3) an attention-control condition that is time-equivalent to condition 2 above, and addresses diet, exercise, and HIV. Thus we will determine whether longer-term maintenance of safer sex behaviors is possible among HIV+ methamphetamine-using MSM, a population that remains at very high risk of HIV transmission, and for which substitution therapies to promote cessation and risk reduction are not yet available.

ELIGIBILITY:
Inclusion Criteria:

* HIV+
* Used methamphetamine at least twice in last two months
* At least some recent sexual partners were male
* At least some recent sexual activity has been high-risk for transmission of HIV

Exclusion Criteria:

* Current major psychiatric diagnosis
* Only HIV+ sex partners in past two months
* Consistently protected sex with HIV- or serostatus-unknown partners in last two months
* Sexually inactive in last two months
* Found out about HIV+ status less than two months ago

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 429 (Actual)
Dates: Start 2007-02; Primary Completion 2012-04 (Actual); Study Completion 2012-04 (Actual)

PRIMARY OUTCOMES:
Reduction of defined sexual risk behaviors | 18 months

CONTACTS AND LOCATIONS:
Overall Officials: Thomas L. Patterson, Ph.D., Principal Investigator — University of California, San Diego
Locations (1):
- Webster Building, 3500 Fifth Ave., Suite 102, San Diego, California, United States

REFERENCES:
- [Derived] Semple SJ, Strathdee SA, Zians J, Patterson TL. Factors associated with sex in the context of methamphetamine use in different sexual venues among HIV-positive men who have sex with men. BMC Public Health. 2010 Apr 1;10:178. doi: 10.1186/1471-2458-10-178. PMID 20359362